CLINICAL TRIAL: NCT03012737
Title: Palliation of Dyspnea With Mouth Piece Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in finding suitable patients.
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Lauri Lehtimäki, Associate professor, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R16111
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MPV arm (Other): Subjects use mouth piece ventilation (MPV) accoring to their will to alleviate dyspnea for 24 hours.
  Interventions: Device: Trilogy 100 ® (Philips Respironics)

INTERVENTIONS:
Device: Trilogy 100 ® (Philips Respironics) — Trilogy 100 ® (Philips Respironics) on MPV mode.
  Other Names: Mouth piece ventilation

SUMMARY:
An uncontrolled feasibility study on using mouth piece ventilation in palliation of dyspnea in subjects with incurable advanced disease. Subjects are recruited from a local Hospice and from oncology ward. The main outcomes are the compliance of the subjects with the treatment and alleviation of dyspnea during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* at least moderate dyspnea (NRS = Numeric Rating Scale ≥ 4)
* incurable advanced disease
* able to understand the study and to give informed consent
* would not gain from intensive care or resuscitation according to the treating physician

Exclusion Criteria:

* unable to participate and use MPV due to e.g. delirium or lack of co-operation
* the cause of the dyspnea can be succesfully treated
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in dyspnea after initial use of MPV | 5 - 60 min

SECONDARY OUTCOMES:
Change in dyspnea after 24 hours of using MPV | 24 hours
Proportion of subjects having side-effects or not being compliant with MPV | 24 hours
Proportion of subjects gaining from MPV | 24 hours
Proportion of subjects willing to continue on MPV after the intervention | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Lehtimäki, MD, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - Dpt of oncology, Tampere University Hospital, Tampere
  - Pirkanmaa Hospice, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lehto JT, Leivo-Korpela S, Korhonen T, Rantala HA, Raunio H, Lyly-Yrjanainen T, Lehtimaki L. Mouthpiece ventilation in the management of dyspnea: A single-arm pilot study. Palliat Med. 2020 Oct;34(9):1274-1278. doi: 10.1177/0269216320935003. Epub 2020 Jun 24. PMID 32579086